CLINICAL TRIAL: NCT02049606
Title: Double Blinded, Randomized, Active Drug Comparative, Multi-center, Phase Ⅳ Clinical Study to Compare the Efficacy and Safety of LAYLA in Osteoarthritis Patients of the Knee.
Brief Title: To Compare the Efficacy and Safety of LAYLA in Osteoarthritis Patients of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PMG Pharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAYLA_P4_NB
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: LAYLA; Non-inferiority; 100mm pain VAS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Nabumetone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAYLA (Experimental): Drug : LAYLA tablet/bid
  Interventions: Drug: LAYLA tablet
- CENATONE (Active Comparator): Drug : CENATONE tablet/qd
  Interventions: Drug: CENATONE tablet

INTERVENTIONS:
Drug: LAYLA tablet — 1 Tablet twice a day
  Other Names: LAYLA 405.4mg
  Arms: LAYLA
Drug: CENATONE tablet — 2 Tablets once a day
  Other Names: Nabumetone 500mg
  Arms: CENATONE

SUMMARY:
This is a randomized, double-blind study to compare the efficacy and safety of LAYLA tablet and CENATONE tablet in the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥40 and ≤80 years of age
* Radiographic evidence of grade 1,2 or 3 osteoarthritis based on the Kellgren & Lawrence radiographic entry criteria
* Stable osteoarthritis during 3 months
* Score of 100mm Pain VAS ≤ 80mm at screening
* Score of 100mm Pain VAS ≥ 40mm at baseline
* Written consent form voluntarily

Exclusion Criteria:

* Disease of spine or other Lower limb joints that could affect fo evaluate the efficacy
* History of surgery or arthroscopy of the study joint within 6 months
* Trauma of study joint within 12 months
* Medication of constantly(more than 1 week) corticosteroid by oral within 3 months
* Diagnosed with psychical disorder, and taking medication
* Medication of intra-articular injection within 3 months
* Uncontrollable Hypertension patients at screening test
* History of upper gastrointestinal ulceration within 6 months, History of upper gastrointestinal bleeding within 12 months
* History of lower gastrointestinal bleeding within 12 months
* History of coronary artery bypass, systemic lupus erythematosus or mixed connective tissue disease
* Serum creatinine, ALT, AST, total bilirubin over ULN X 2.0 at screening test
* History of hypersensitivity of LAYLA, CENATONE or NSAIDs
* Participation in another clinical trials within 4 weeks
* Medication of constantly (more than 1 week) narcotic analgesics within 3 months
* Not consent about using effectual contraception method during trial
* Pregnant or lactating woman
* History of malignant tumor within 5 years
* Investigator's judgment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Changes from the baseline in 100mm Pain VAS | Baseline through week8

SECONDARY OUTCOMES:
Changes rate from the baseline in 100mm Pain VAS | 8 weeks
Changes from the baseline in WOMAC | 8 Weeks
Changes from the baseline in EQ-5D | 8 Weeks
Changes in the patient self-assessed overall symptom score | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seung Baik Kang, MD, Principal Investigator — SMG-SNU Boramae Medical Center; Jeong Ku Ha, MD, Principal Investigator — Inje University; Han Jun Lee, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Yong In, MD, Principal Investigator — The Catholic University of Korea; Jong Min Kim, MD, Principal Investigator — Asan Medical Center; Sahng Hoon Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul